CLINICAL TRIAL: NCT00584857
Title: A Phase II Study of Combination Therapy With Paclitaxel, Carboplatin and Megesterol Acetate for the Management of Advanced Stage or Recurrent Carcinoma of the Endometrium
Brief Title: A Phase II Study of Therapy With Paclitaxel, Carboplatin and Megesterol Acetate for the Management of Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, J. Michael Straughn, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F040628007 (UAB 0403); UAB 0403 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Single
  Interventions: Drug: Paclitaxel ,Carboplatin , Megesterol Acetate

INTERVENTIONS:
Drug: Paclitaxel ,Carboplatin , Megesterol Acetate — Paclitaxel will be administered at an appropriate dose (175mg/m2) as a 3 hour continuous IV infusion every 21 days. Carboplatin will be administered at an appropriate dose utilizing Calvert formula for determining the area under the curve (AUC) based on the patient's glomerular filtration rate. Megesterol Acetate will be given orally four times a day at an anti-tumor dosage of 40 mg. This will be given for a total of 6 cycles over 18 weeks with the Megace continuing for 5 years as long as no evidence of recurrence is present.

SUMMARY:
This is a study to determine the optimal treatment for patients with advanced stage or recurrent endometrial cancer. Traditionally, patients have been treated with either hormonal therapies (megesterol) or chemotherapy (paclitaxel and carboplatin). This study investigates the effectiveness of the combination of hormonal therapy and chemotherapy. This study also will examine the side-effects associated with these drugs and the quality of life of patients on combination therapy.

DETAILED DESCRIPTION:
Endometrial cancer is the most common gynecologic malignancy with 40,100 new cases diagnosed and 6,800 deaths attributable to this malignancy in 2003. Most patients diagnosed with endometrial cancer have early stage disease that is amenable to treatment with hysterectomy and bilateral salpingo-oophorectomy with excellent clinical outcomes. Surgical staging has improved accuracy over clinical staging for defining a low risk population of patients who have favorable long-term outcomes with surgery alone. However, approximately 15% of patients will have evidence of Stage III or IV disease at the time of initial diagnosis and 15% of surgical Stage I/II patients will have recurrent disease. Radiation therapy will be effective in patients with disease confined to the pelvis; however, patients with metastatic disease will require more systemic therapy in order to control disease.

Multiple chemotherapeutic agents including cisplatin, doxorubicin HCL, paclitaxel, carboplatin, and oral etoposide, alone and in combination, have been studied for persistent, advanced or recurrent endometrial cancer. A phase III study by the Gynecologic Oncology Group (GOG) compared doxorubicin with and without cisplatin (GOG 107) for patients with advanced or recurrent endometrial cancer. A higher response rate (45% vs. 27%) was noted for combination therapy and has been considered by many to be the standard chemotherapy regimen for treatment of patients with advanced endometrial cancer. However, clinical trials have continued to define the optimal chemotherapy regimen for this disease. Recently, the use of whole abdominal radiation therapy in the adjuvant setting for advanced endometrial cancer was demonstrated to be inferior to the combination of cisplatin and doxorubicin. The predicted 2-year survival of 70% for patients receiving the chemotherapeutic regimen was superior to patients that received radiation therapy (59%)(p<0.01).

Hormonal and cytotoxic chemotherapy agents are utilized in patients with metastatic or recurrent disease not amenable to radiation therapy. Hormonal agents have been used in this disease process since it has been demonstrated to be a hormonal responsive tumor. Notably, a correlation between histologic grade and the presence or absence of hormonal receptors has been noted, with well differentiated tumors more likely to express hormone receptors than those with poor histology. Furthermore, the presence of estrogen receptors (ER) and progesterone receptors (PR) varies with tumor histology. ER has been reported to be present between 70% and 87% of endometrioid adenocarcinoma and 0 and 24% in UPSC; while, PR has ranged from 67% to 91% in endometrioid tumors and 0 and 19% in UPSC.

Various progestins have been investigated including Megace (megesterol acetate) and Provera (medroxyprogesterone acetate) for the treatment of endometrial cancer. These agents are generally well tolerated and have been reported to have response rates of 15-30% with long-term complete responses not uncommonly experienced. Furthermore, median survival in patients treated with progestins ranges from 9 to 20 months.

As paclitaxel has been noted to be active in ovarian cancer and other malignancies, it seems reasonable to evaluate its utility for endometrial cancer. Accordingly, single agent paclitaxel was administered to 30 chemotherapy naïve patients with advanced or recurrent endometrial cancer. The overall response rate was 36% when patients received a 24-hour infusion of paclitaxel. Furthermore, paclitaxel given as a 3-hour infusion demonstrated a response between 27 to 37% in patients that had failed prior chemotherapy.

Paclitaxel has been combined with platinum compounds, primarily cisplatin in several studies. A phase II study that combined paclitaxel 175 mg/m2 as a 3-hour infusion with cisplatin 75 mg/m2 reported a 67% response rate. There were seven complete responses and nine partial responses with an 18 month median overall survival. An additional phase II study evaluated the efficacy of combining paclitaxel and carboplatin in both primary advanced and recurrent non-papillary and papillary tumors following radiation. The response rate was 78% in patients with primary advanced non-papillary tumors with a median disease-free survival of 23 months, with the median overall survival not being reached at the time of publication. Furthermore, patients with recurrent endometrial cancer had a response rate of 56%, with a median overall survival of 15 months.

A phase I study by the GOG combined paclitaxel, cisplatin, and doxorubicin with or without granulocyte colony-stimulating factor. A 46% response rate with this regimen determined the optimal dosing of the agents and led to a phase III GOG study (GOG 177). GOG 177 demonstrated the combination of paclitaxel, doxorubicin and cisplatin to have higher response rates (57% vs. 33%) over the combination of doxorubicin and cisplatin, but the three drug combination was associated with more toxicity and 12-month overall survival (58% vs. 50%) was similar. Furthermore, more Grade 3 and 4 toxicity was experienced by patients that received the three drug combination, although this was not statistically significant. Accordingly, a phase III trial comparing the paclitaxel, doxorubicin, and cisplatin regimen to a more tolerable regimen of paclitaxel and carboplatin is planned by the GOG, based on equivalency studies in ovarian cancer patients where carboplatin was substituted for cisplatin and demonstrated easier administration with equal efficacy and less toxicity.

The combination of hormonal agents with cytotoxic chemotherapy has also been investigated. These studies utilized various combinations of non-taxane based cytotoxic chemotherapy in addition to megesterol or medroxyprogesterone acetate. Patients had response rates that varied from 33% to 60%, with the combination cyclophosphamide, doxorubicin, cisplatin and megesterol producing the greatest response rate. Additionally, Pinelli et al. reported a 56% complete or partial response rate in a group of patients treated with carboplatin and sequential hormonal therapy with megesterol and tamoxifen. These studies suggest that sequential administration of hormonal therapy with chemotherapy has no detrimental effects on patients, and may be beneficial as hormonal therapy is generally less toxic than chemotherapy. Based on known tolerability and efficacy, investigating the combination of megesterol acetate with paclitaxel and carboplatin chemotherapy appears to be a reasonable option in the setting of advanced or recurrent endometrial cancer.

Accordingly, this phase II study will evaluate the combination of paclitaxel, carboplatin and megesterol acetate for the treatment of advanced or recurrent adenocarcinoma of the endometrium.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy proven endometrioid adenocarcinoma or adenosquamous carcinoma.
* Patients must have evidence of primary FIGO Stage III-IVB or recurrent endometrial cancer.
* Patients with non-measurable disease following complete cytoreduction at the time of initial operative management for Stage III-IVB are eligible.
* Patients with recurrent disease must have disease confirmed by one of the following:

  1. CT Scan
  2. MRI
  3. PET Scan
  4. Physical Exam
* Patients must have adequate organ function defined as:

  1. Platelets >/= 100,000/1
  2. Granulocytes (ANC) >/= 1,500/
  3. Creatinine </= 1.6mg/dl
  4. SGOT (AST) </= 3x upper limits of normal
  5. Bilirubin within institutional normal limits
* Patients must have adequate performance status (ECOG performance status 0-2.
* Patients must be age 19 or greater and have signed informed consent.

Exclusion Criteria:

* Patients with history of other malignancies (except non-melanoma skin cancer or carcinoma-in-situ of the cervix) are ineligible.
* Patients with high-risk histologic subtypes of endometrial cancer, namely papillary serous or clear cell histology are ineligible.
* Patients with evidence of uterine sarcoma, including leiomyosarcoma, carcinosarcoma, endometrial stromal sarcoma, and adenosarcoma are ineligible.
* Patients who are less than 8 weeks after the completion of radiotherapy are ineligible.
* Patients receiving any other investigational agents are ineligible.
* Patients with known hypersensitivity to paclitaxel, carboplatin, or megesterol are ineligible.
* Patients with uncontrolled current illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, serious peripheral neuropathy, or psychiatric illness/social situations that would limit or preclude compliance with study requirements are ineligible.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Straughn, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Women's and Infant Center, 1700 6th Ave S, Birmingham, Alabama, United States

REFERENCES:
- [Result] Bevis KS, Kilgore LC, Alvarez RD, Straughn JM Jr, Leath CA 3rd. Combination therapy with paclitaxel, carboplatin and megestrol acetate for the management of advanced stage or recurrent carcinoma of the endometrium: a phase II study. J Reprod Med. 2014 Mar-Apr;59(3-4):113-20. PMID 24724218

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel/Carboplatin/Megesterol Acetate: Paclitaxel will be administered at 175mg/m2) as a 3 hour continuous IV infusion every 21 days. Carboplatin will be administered at a dose utilizing Calvert formula for determining the area under the curve (AUC) based on the patient's glomerular filtration rate. Megesterol Acetate will be given orally four times a day at a dosage of 40 mg.
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin/Megesterol Acetate
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel/Carboplatin/Megesterol Acetate
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival
Description: Number of subjects alive at 3 years
Time Frame: 3 years - median followup of 40.4 months
Measure: Number; unit: partipants
Arm/Group | Paclitaxel/Carboplatin/Megesterol Acetate
Number analyzed (Participants) | 28
partipants | 17

2. Secondary Outcome: Toxicity
Description: Toxicity secondary to paclitaxel, carboplatin, and megesterol acetate based on NCI common toxicity criteria
Time Frame: 3 years
Measure: Number; unit: participants
Arm/Group | Paclitaxel/Carboplatin/Megesterol Acetate
Number analyzed (Participants) | 30
participants | 5

ADVERSE EVENTS:
Arm/Group | Paclitaxel/Carboplatin/Megesterol Acetate
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel/Carboplatin/Megesterol Acetate (N=30)
deep vein thrombosis (Vascular disorders) | 3 (3)
port fracture (Surgical and medical procedures) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes